CLINICAL TRIAL: NCT01474408
Title: Venous Function in Cardiovascular Disease Patients; The Neglected Part of Circulatory Regulation
Brief Title: Venous Function in Cardiovascular Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/760
Record Dates: First submitted 2011-11-04; First posted 2011-11-18 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Myocardial Infarction
Keywords: Coronary artery bypass; Exercise therapy; Revascularization (PCI)
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- interval training (Experimental): 4 x 4 minutes exercise at 90 - 95 % of peak heart rate separated with 3 minutes at 70 % of peaks heart rate
  Interventions: Behavioral: interval training day 1; Behavioral: Moderate exercise day 2; Behavioral: Control day 3
- moderate exercise (Active Comparator): moderate continuous exercise at 70 % of peak heart rate on venous function.
  Interventions: Behavioral: interval training day 1; Behavioral: Moderate exercise day 2; Behavioral: Control day 3
- control (Other): routine measurements, no exercise
  Interventions: Behavioral: interval training day 1; Behavioral: Moderate exercise day 2; Behavioral: Control day 3

INTERVENTIONS:
Behavioral: interval training day 1
  Other Names: aerobic interval training
Behavioral: Moderate exercise day 2
Behavioral: Control day 3

SUMMARY:
The primary aim is to determine the acute effect of two different training interventions on venous plasticity in patients with myocardial infarction (MI), revascularization or coronary artery graft surgery compared to age-matched healthy subjects.

DETAILED DESCRIPTION:
Compare the effect of 4 x 4 minutes at 90 - 95 % of peak heart rate separated with 3 minutes at 70 % of peaks heart rate and moderate continuous exercise at 70 % of peak heart rate on venous function.

ELIGIBILITY:
Inclusion Criteria:

* myocardial infraction (MI)
* revascularization (PCI)
* coronary artery bypass graft surgery (CABG)

Exclusion Criteria:

* unstable angina pectoris
* uncontrolled hypertension
* orthopedic and/or neurological limitations
* participation in other studies
* MI (closer than 4 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Venous Compliance change | 48 hours
  Measured by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- Institutt for Sirkulasjon og Bildetechnikk, NTNU, Trondheim, Norway

REFERENCES:
- [Result] Leinan IM, Aamot IL, Stoylen A, Karlsen T, Wisloff U. Upper arm venous compliance and fitness in stable coronary artery disease patients and healthy controls. Clin Physiol Funct Imaging. 2017 Sep;37(5):498-506. doi: 10.1111/cpf.12324. Epub 2015 Dec 15. PMID 26667796